CLINICAL TRIAL: NCT00820183
Title: A Quality Improvement Plan for Hypertension Control: the INCOTECA Project
Brief Title: A Quality Improvement Plan for Hypertension Control
Acronym: INCOTECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Roser VallésFernández, Institut Català de la Salut
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RSB_2006
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension
Keywords: Hypertension; Intervention; Primary Care; Quality improvement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- quality improvement plan (Experimental): It will be the group of primary health care teams who will undertake the quality improvement plan for hypertensive patients
  Interventions: Other: Quality Improvement plan for Hypertension Control
- non intervention (No Intervention): It will be the group of primary health care teams that will not undertake the quality improvement plan for hypertension control

INTERVENTIONS:
Other: Quality Improvement plan for Hypertension Control — Implementation of a plan of quality improvement addressed to health professionals in Primary Health Care Teams. It includes:
  Specific training programme on how to diagnose hypertension , and measure blood pressure correctly To send feed back information to primary care health professionals about poorly controlled hypertensive patients An audit will be performed, every 6 months, to see the adhesion to the recommended clinical guidelines , and the information will be diffused among the participant primary health care professionals Each participant primary health care team will have a designated reference person, that will provide support on any doubts on the programme implementation
  Arms: quality improvement plan

SUMMARY:
The study hypothesis is that the implementation of a plan for quality improvement at the primary care health teams taking care of hypertensive patients, will increase the level of blood pressure control among those patients.

DETAILED DESCRIPTION:
The study is to compare the results on the hypertension control between two groups of primary health care teams. The intervention group will undertake a quality improvement plan for hypertension control, in which the following aspects will be included in the intervention:

Specific training programme on how to diagnose hypertension , and measure blood pressure correctly To send feed back information to primary care health professionals about poorly controlled hypertensive patients An audit will be performed, every 6 months, to see the adhesion to the recommended clinical guidelines , and the information will be diffused among the participant primary health care professionals Each participant primary health care team will have a designated reference person, that will provide support on any doubts on the programme implementation.

The non intervention group will follow hypertensive patients following the same clinical practice guide as the intervention group, with no intervention on the primary health care professionals

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hypertension before January 1st, 2006
* Patients assigned at the primary health team participating, and with clinical electronic records

Exclusion Criteria:

* Patients diagnosed with hypertension after January 1st, 2006
* Patients under 18 years of age
* Patients with a diastolic blood pressure higher than systolic blood pressure as recorded in the clinical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34327 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
good control of hypertension as a dichotomous variable, based on systolic blood pressure and diastolic blood pressure records over the last 12 months | every three months, for a whole year

SECONDARY OUTCOMES:
treatment with antihypertensive drugs, number of antihypertensive drugs, assessment of therapeutic compliance | every three months, for a whole year

CONTACTS AND LOCATIONS:
Overall Officials: Roser Valles Fernandez, Principal Investigator — Institut Català de la Salut
Locations (1):
- SAP Cerdanyola-Ripollet Institut Català de la Salut, Cerdanyola del Vallès, Barcelona, Spain

REFERENCES:
- See also: describes de procedures to follow management and treatment of hypertensive patients in the study protocol — http://www.gencat.cat/ics/professionals/guies/hipertensio/hipertensio.htm